CLINICAL TRIAL: NCT06910787
Title: Outpatient Virtual Reality-Directed Treatment for Pain in Inflammatory Bowel Disease
Brief Title: Outpatient VR (Virtual Reality)-Brain-gut Behavioral Therapies (BGBT) in Inflammatory Bowel Disease (IBD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American Gastroenterological Association (Other)
Responsible Party: Principal Investigator, Shirley Cohen-Mekelburg, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00267700
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Virtual Reality; Outpatient; Pain; Brain Gut Behavioral Treatment; Enhanced treatment as usual; Randomized
MeSH Terms: conditions — Inflammatory Bowel Diseases; Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to Enhanced Treatment as Usual (E-TAU) or VR-directed BGBT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- VR-directed BGBT (Experimental)
  Interventions: Device: VR-directed BGBT
- Enhanced treatment as usual (E-TAU) (Active Comparator)
  Interventions: Other: E-TAU

INTERVENTIONS:
Device: VR-directed BGBT — VR-directed BGBT using the Oculus Meta Quest 3 VR headset will be delivered using the Synergi application. The program includes 4-weeks of daily self-led activities using 5 virtual modules: (1) education (2) two interactive games (3) breathing exercises (4) gut-directed meditation and (5) gastroenterology-specific Cognitive behavioral therapy (CBT). Participants will also receive standard care. On day 1, intervention arm participants will undergo a brief in-person or virtual (i.e., zoom or Microsoft teams) training with study staff to learn how to use the VR headset and access intervention modules. On day 1 participants will be asked to explore each of the program modules to achieve initial familiarity. Participants will be encouraged to use the VR-BGBT program for at least 15 minutes daily, but at minimum 3-4 days each week. Additionally, study assessments will be completed at baseline, 2-weeks, 4-weeks, and 8-weeks, with an interview within 1-2 weeks of completing the program.
  Arms: VR-directed BGBT
Other: E-TAU — Participants will receive standard of care, as directed by the participant's gastroenterologist. Participants will also receive an educational video and fact sheet on pain in IBD. This will be 4-weeks with study assessments at baseline, 2-weeks, and 4-weeks, 8-weeks.
  Arms: Enhanced treatment as usual (E-TAU)

SUMMARY:
This research study is being done to learn if a virtual reality (VR)-directed BGBT program is feasible and acceptable for patients to enhance pain treatment for patients with IBD.

The study hypothesis include:

* the study will achieve greater than 75% program completion and 75% study assessment completion
* patients with IBD will find VR-directed BGBT acceptable as an outpatient pain treatment
* outpatient VR-directed BGBT in IBD arm participants will report a greater reduction in pain scores, symptom burden, stress, depression, anxiety, and pain-related interference and an improvement in health-related quality of life
* will have lower opioid requirements and healthcare utilization at 4-weeks follow-up compared to the E-TAU arm

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients (18 years and older) that carry a diagnosis of IBD and confirmed in the electronic health record (EHR) as receiving IBD-targeted treatment
* IBD-targeted treatment include 5-aminosalicylates, thiopurines, biologics, or small molecules such as Janus kinase inhibitor (JAK) inhibitors or sphingosine-1-receptor modulators.
* Self-report abdominal pain with an average severity ≥ 2 on a 0-10 pain scale over the last 24 hours,
* Participants are willing and able to pick-up and drop-off VR equipment at University of Michigan (UM)

Exclusion Criteria:

* Patients that do not report pain (i.e., score<2) as they are less likely to benefit from VR-directed BGBT
* Patients with a history of conditions that could potentially be harmed by VR including seizures/epilepsy, loss of awareness, binocular vision loss, current pregnancy, or uncontrolled cardiac (e.g., arrhythmia, coronary artery disease) or neurological/cerebrovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility defined by the proportion of enrolled participants that complete the 4-week VR-directed BGBT program and study assessments. | 4 weeks
  The study team hypothesizes the study will achieve greater than 75% program completion and 75% study assessment completion.
Acceptability of VR-directed BGBT based on a semi-structured post intervention interview | 4 weeks
  The interview will be done to understand the participants' experience with the VR-directed BGBT intervention and conducted using interview guides with open-ended questions. interview guides will focus on four main domains related to participant's pain history, experience with VR-directed BGBT (including tolerability and acceptability of each BGBT module), perceived impact (including information on any components that were perceived to be most helpful or ineffective), and suggested improvements for program refinement.
VR-BGBT acceptability using the Treatment Acceptability and Adherence Scale | 4 weeks
  This is a 10-question scale that participants choose from 1 (disagree strongly) - 7 (agree strongly). Scores range from 10-70 with higher scores indication greater acceptability.
VR-BGBT usability using the System Usability Scale | 4 weeks
  This is a 10-question scale that participants choose from 1 (strongly agree) - 5 (strongly disagree). Scores range from 0 to 100 with a higher score indicating greater acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Cohen-Mekelburg, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No